CLINICAL TRIAL: NCT01569698
Title: Modalities of Renal Replacement Therapy in Pediatric Acute Kidney Injury
Acronym: EPURE
Status: Terminated | Type: Observational
Why Stopped: sponsor and investigator's decision
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-A00670-39
Record Dates: First submitted 2012-03-23; First posted 2012-04-03 (Estimated); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Kidney Failure, Acute
Keywords: pediatric; acute renal failure; acute extra renal replacement therapy; Intermittent Hemodialysis; Continuous Renal Replacement Therapies; Peritoneal Dialysis
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- extrarenal replacement therapy: Intermittent Hemodialysis, Continuous Renal Replacement Therapies, and Peritoneal Dialysis
  Interventions: Procedure: acute extra renal replacement therapy

INTERVENTIONS:
Procedure: acute extra renal replacement therapy — usual modalities of pediatric acute extra renal replacement therapy : Intermittent Hemodialysis, Continuous Renal Replacement Therapies, and Peritoneal Dialysis
  Other Names: Non applicable.

SUMMARY:
Limited prospective data is available to compare morbidity and mortality between renal replacement modalities in pediatric acute renal failure.

In the absence of clear standard of care, the choice of the extra renal replacement therapy modality is subject to clinical judgement, practical aspects, and costs.

This study will supply important data about usual modalities of pediatric acute extra renal replacement therapy and their impact on patient outcome and renal recovery. An obvious next step will be to conduct a randomized controlled trial comparing the different strategies.

DETAILED DESCRIPTION:
In children, there are limited data on extra renal replacement therapy. Pediatric studies are often retrospective, or often limited to specific disease processes or specific extra renal therapy. The lack of large studies including different usual modalities in pediatrics limits any formal recommendation on use in relation to patient outcomes, including renal recovery and mortality. Some of the issues that need consideration are the choice of dialysis modality (including Intermittent Hemodialysis, Continuous Renal Replacement Therapies, and Peritoneal Dialysis), the indications for and timing of dialysis intervention, the dose of dialysis and their effects on outcomes from acute kidney injury in children.

This study will supply important data about pediatric acute extra renal replacement therapy, including the epidemiology of pediatric acute kidney injury leading to extra renal replacement therapy, the variety of the treatment modalities, and their effects on the course of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years, including the newborn ;
* Acute kidney injury as defined by pRIFLE classification requiring extra renal replacement therapy, whatever is the method.

Exclusion Criteria:

* Treatment by extra renal replacement therapy for terminal renal failure;
* History of renal transplantation;
* Extra renal replacement therapy for an inborn errors of metabolism without acute renal failure;
* Extra renal replacement therapy in the context of a drug intoxication without acute renal failure;
* Treatment by technique in MARS (Molecular Adsorbent Recirculating System);
* Modified ultrafiltration during surgery.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with an acute renal failure
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2012-06; Primary Completion 2016-11 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
extra renal replacement therapy | at day 60 +/- 7
  To describe usual modalities of pediatric acute extra renal replacement therapy including Intermittent Hemodialysis, Continuous Renal Replacement Therapies, and Peritoneal Dialysis.

SECONDARY OUTCOMES:
Current incidence | at day 60 +/- 7
  Current incidence of the use of extra renal replacement therapy in pediatric acute renal failure
etiologies | at day 0
  Acute kidney injury etiologies leading to extra renal replacement therapy
Risk factors of mortality and non recovery of the renal function | at day 60
  Risk factors of mortality and non recovery of the renal function at day 60 in child acute kidney injur treated by extra renal replacement therapy (including, among others, the choice of dialysis modality (i.e. Intermittent Hemodialysis, Continuous Renal Replacement Therapies, and Peritoneal Dialysis), the indications for and timing of dialysis intervention, and the dose of dialysis).
  Urea, blood pressure, creatinine, report proteinuria / creatinuria, renal disease, acute graft

CONTACTS AND LOCATIONS:
Overall Officials: Theophile Gaillot, MD, Principal Investigator — Rennes University Hospital
Locations (19):
- Canada (2):
  - Pediatric intensive care - Centre mère enfants, Sainte-Foy
  - Pediatric intensive care -, Sherbrooke
- France (16):
  - Angers University Hospital, Angers
  - Besançon University Hospital, Besançon
  - Pediatry - Bordeaux University Hospital, Bordeaux
  - Reanimation pediatric - Morvan Hospital, Brest
  - Pediatry - Cote De Nacre University Hospital, Caen
  - Pediatric nephrology - Hôpital Couple-enfants, Grenoble
  - Bicêtre University Hospital, Le Kremlin-Bicêtre
  - Pediatry - Hopital de la Mère et de l'Enfant, Limoges
  - Anesthesy-Pediatric reanimation - Nord University Hospital, Marseille
  - Pediatric Nephrology and dianetology - Arnaud de Villeneuve Hospital, Montpellier
  - Pediatric reanimation - Hôpital mère-enfant, Nantes
  - Réanimation et Surveillance - Robert Debre Hospital, Paris
  - Pediatry - Reims University Hospital, Reims
  - Nephrology - Hôpital des enfants, Toulouse
  - Nephrology - Pediatric emergency - Clocheville University Hospital, Tours
  - Pediatric reanimation - Brabois Hospital, Vandœuvre-lès-Nancy
- Groupe hospitalier Sud Reunion, Réunion, Reunion